CLINICAL TRIAL: NCT06161324
Title: The Effectiveness of a Tele-rehabilitation Program Implemented in a Greek Clinical Setting for Women With Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Tele-rehabilitation for Women With Urinary Incontinence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Evdokia Billis, Professor in Physiotherapy, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Telerehab and incontinence
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Urinary Incontinence
Keywords: Tele-rehabilitation; urinary incontinence; stress incontinence; pelvic floor muscle exercise; adherence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will remain hidden from the responsible physical therapist who will implement the treatment in the groups (he/she will be informed on the first day of the intervention for each patient). Due to the nature of the treatment, the intervention is not blinded between participants and clinicians. However, the analysis of the data will be 'blind' to all both parties, assessor and investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tele-rehabilitation group (TeleG) (Experimental): The participants of the tele-rehabilitation group(TeleG), will remotely perform a pelvic floor muscle (PFM) exercises program at home in cooperation with a PFM superficial sensor. At the same time, the participants will be supervised remotely by the physiotherapist. Participants and therapist will communicate through the mobile app, either synchronously (i.e. through video calls) or asynchronously (i.e. through emails), regarding the execution of the PFM exercises (direction of the PFM contraction, frequency of the PFM exercise program etc.)
  Interventions: Other: PFM exercises program through the Mobile app in cooperation with the superficial sensor
- Traditional treatment group (TrG) (Active Comparator): In the Traditional (classic) treatment group (TrG), participants will follow the usual care treatment of pelvic floor muscles, based on the "pragmatic" treatment of urinary incontinence, which is used today in rehabilitation clinics, centers etc.
  Interventions: Other: Face-to face PFM exercises program in Healthcare environment
- Control Group (CG) (Other): The participants of the control group (CG), will follow a pelvic floor muscle exercise program at home (via leaflet), without any supervision.
  Interventions: Other: PFM exercises program via home-leaflet(without suprevision)

INTERVENTIONS:
Other: PFM exercises program through the Mobile app in cooperation with the superficial sensor — The mobile app will offer a personalized progressive protocol to the user based on his needs, via 12 levels of games(from the easiest to the hardest).The cooperating PFM superficial sensor will indicate the activity of the PFMs during the contraction.Νο face-to-face meetings will be incurred between participants and therapist.
  Participants will follow a program for 12 weeks(3 times weekly, 1-5 sessions daily, each session's duration approximately 20 minutes).Endurance training will involve slow velocity contraction and speed training will involve quick (i.e.1 sec duration) strong contractions."Knack maneuver" training will contain a pre-contraction before the increment of the intra-abdominal pressure during coughing. The exercise positions will change every 2 weeks (supine, side, prone, quadruped support, sitting and standing position).
  Arms: Tele-rehabilitation group (TeleG)
Other: Face-to face PFM exercises program in Healthcare environment — The therapy will include face-to-face meetings weekly, regarding the progress of the treatment and its smooth transition (intra-vaginally assessment when it needs, correction, encouragement, motivation, etc).
  Participants will follow a personalized progressive PFM exercise program for 12 weeks (3 times weekly, 1-5 sessions daily, each session's duration approximately 20 minutes).The endurance training will involve slow velocity contraction and the speed training will involve quick (i.e.1 sec duration) strong contractions. The "Knack maneuver" training will contain a pre-contraction before the increment of the intra-abdominal pressure during coughing. The exercise positions will change every 2 weeks.It will be followed the order of supine, side, prone, quadruped support, sitting and standing position
  Arms: Traditional treatment group (TrG)
Other: PFM exercises program via home-leaflet(without suprevision) — The participants of the CG will be advised to follow a personalized PFM exercise program at home based on their 1st meeting assessment. They will receive a comprehensive leaflet, with instructions and images about the PFM exercises at home. The PFM exercise program will last 12 weeks (3 times weekly, 1-5 sessions daily), without meetings, guidance and supervision by the physiotherapist. Similarly to the other two intervention groups, the program will contain endurance training (slow velocity contraction), speed training (quick contractions), "Knack maneuver" training (pre-contraction before coughing), and changing positions every 2 weeks (supine, side, prone, quadruped support, sitting and standing position)
  Arms: Control Group (CG)

SUMMARY:
The prevalence of urinary incontinence (UI) in the female Greek population is 1 to 3 women (27%).Globally, the development of tele-rehabilitation programs through mobile application (mobile apps) has been a breakthrough for UI treatment. More specifically, the pelvic floor muscles (PFM) exercise programs through mobile apps, provide optimal health care services by offering to the patients a therapy program in the convenient environment of their choice (e.g their homes), with safety and less expense. Furthermore, it is given the opportunity to patients with mobility problems or with lack of transport or to them who live in remote areas, to treat their incontinence.

However, the majority of the existence mobile apps, work as simple verbal instructions and they do not being tailored in patients' individual needs, which is necessary for the successful implementation of the PFM exercise programs. Additionally, the PFM training is effective for UI treatment, when occurs intensively (daily) with supervision for at least 3 months by a physiotherapist. However, the adherence to a such intensive treatment program is very often compromised, because of many reasons (e.g lack of interest etc).

Therefore the main purpose of the current study is, to investigate the effectiveness of a tele-rehabilitation program, through a novel, innovative mobile app (customized in patients needs), in cooperation with a PFM superficial sensor. The mobile app will offer an interactive environment and the opportunity of a simultaneous supervision by a physiotherapist during the treatment, which might provide sufficient motivation to the patient to adhere with the intensive PFM exercise program. A secondary objective of the study is, to investigate the degree of adherence to PFM exercises and the degree of supervision, which is needed in the tele-rehabilitation program. Both the mobile app and the PFM superficial sensor, will be created for the needs of the present study.

DETAILED DESCRIPTION:
The present study is designed to be conducted as a prospective randomized controlled clinical trial (RCT) with three arms.

1. The Telerehabilitation Group (TeleG) will use the mobile app in collaboration with the pelvic floor muscle (PFM) superficial sensor, with the remote supervision of the physiotherapist, which will take place in home.
2. Traditional treatment Group (TrG) will follow PFM exercises program with the physiotherapist, which will take place in a health care environment.
3. Control Group (CG) will execute the PFM exercises via a home leaflet, without any supervision.

Αll patients will be assessed in three sessions, at baseline (0 wk), half-way at 6 wks and at the end of the treatment (after 12 wks).

Primary outcome measures will evaluate the severity of the incontinence and the quantity of the urinary loss through the patient-centered International Consultation on Incontinence Questionnaire Short Form (ICIQ-UI-SF) and the clinician-centered '1-hour Pad test', respectively.

Secondary outcomes will include vaginal evaluation through (a) digital palpation using the PERFECT assessment scheme and through (b) an electromyography probe, in order to be assessed the power and the endurance of the PFMs. The patients will complete patient-centered outcome measures, such as a specific PFM exercise adherence questionnaire and a PFM exercise diary during their treatment, in order to be evaluated on how well they followed the program.

Patients will be recruited voluntarily through the University Urology clinic, physician referrals, advertisements in hospitals, posting on the internet, social networks (facebook), etc. Once eligible patients have been selected for treatment, they will fill out an informed consent form.

This study adheres to Ethical considerations and the Helsinki Declaration and is approved by the Research Ethics Committee (R.E.C.) of the University of Patras. All patient data will be stored anonymously/coded in a secure cloud platform accessed only by the research team members. Imputation methods will be applied to address situations where variables are missing, uninterpretable, or inconsistent. Any adverse events will be addressed and documented, while medical consultation will be accessible if needed.

To be ensured the complete allocation concealment of the groups, a randomization process will be used, by a 'blind' researcher who will have no knowledge of the assessment and treatment procedures. The allocation of the participants to the different intervention groups (TeleG, TrG, and CG) will be carried out through a pre-specified computer-generated list, in blocks of six people. Each participant will be randomly assigned a number from the list via a sealed opaque envelope and then the participants will be randomly allocated to the intervention groups via a sealed opaque envelope. To achieve a uniform sample distribution in the intervention groups, each block will include two envelopes for each intervention group (e.g two envelopes for the TeleG, two for the TrG and two for the CG). This method ensures both randomization and concealed allocation, maintaining study integrity and unbiased sample allocation.Due to the nature of the treatment, the intervention is not blinded between participants and clinicians. However, the analysis of the data will be 'blind' (blind-assessor).

It will be performed an analysis based on the data resulting from the initial grouping of patients by treatment protocol (intention-to-treat analysis). The data will be collected in excel tables and through SPSS version 24.0 for Windows and a statistical analysis will be performed. Comparison within the groups before and after the intervention, will be performed by ANOVA using repeated measurements. Comparison between groups after the intervention will be performed by the Student t-test (independent measurements); while the chi-square test will be used for categorical variables (eg yes, no, etc.). In addition, we will calculate the effect size with 95% confidence intervals for each outcome measure with continuous variables. Effect sizes will be considered large if ≥0.8, moderate if ≥0.5 and small if ≥0.2. Results will be considered statistically significant when p<.05. Finally, the results will be presented in means (M) values and their standard deviations (SD).

ELIGIBILITY:
Inclusion Criteria:

* Greek women,
* 18-75 years old,
* Diagnosis of SUI or mixed UI (via Urodynamic test).
* Writing and reading of the Greek language
* Usage of 'smartphones' and internet,
* Able to perform a voluntary muscle contraction of the PFM, during the clinical examination.

Exclusion Criteria:

* 6 months after postpartum,
* Systemic diseases,
* Malignancy,
* Major gynecological surgery (i.e. total hysterectomy) over the last 10 years,
* Neurological dysfunction,
* Mental impairment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on biological gender
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form (ICIQ-UI-SF) | At baseline (0 week), in the middle (6 weeks), and at the end of the intervention (12 weeks)
  Patient-centered questionnaire which contains questions that assess the frequency, severity, and impact of incontinence on patients. The ICIQ-UI SF (range 0-21) is given in four scoring categories: (a) slight symptoms (1-5), (b) moderate symptoms (6-12), (c) severe symptoms (13-18) and (d) very severe symptoms (19-21).
1-hour Pad test | At baseline (0 week) and at the end of the intervention (12 weeks)
  Clinician-centered test by which, the pad is weighed before and after a set of specific-standardized exercises (walking, general exercises, etc.) during one hour. It is compared the difference in the amount of urine retained before and after the exercises in the pad, in order to de determined the urine leakage of the patient.Τhe 1-hour Pad test is given in three scoring categories: (a) mild incontinence (<10 ml) , (b) moderate incontinence (11-50ml) and (c) severe incontinence (>50 ml)

SECONDARY OUTCOMES:
PERFECT assessment scheme | At baseline (0 week), in the middle (6 weeks), and at the end of the intervention (12 weeks)
  Clinician-centered assessment which includes digital intravaginal evaluation of the PFM contraction. The PERFECT assessment scheme, a well recognised and reliable measurement tool for PFMs which evaluates a) the PFMs' power (via Modified Oxford scale) b) the PFMs' endurance in which is recorded the seconds (up to 10 second) that the maximum voluntary contraction (MVC) is held, before a reduction of 50% or more (in power of PFM's) is presented, c) the number of repetitions (up to 10) of the MVC contraction, is held d) the number of fast PFM contractions (up to 10) with one second duration and one second relax, e) the elevation of the posterior vaginal wall, f) the co-contraction with other muscles (like lower abdominals) and g) the involuntary contraction of the PFM on coughing
Electromyographic (EMG) PFM's activity | At baseline (0 week), in the middle (6 weeks), and at the end of the intervention (12 weeks)
  Clinician-centered assessment which includes intravaginal evaluation of the PFM contraction. The intravaginal probe detects the PFMs electromyographic (EMG) activity contraction and presents it in the screen of the computer as a feedback (NeuroTrac® PC Software). Specific PFMs' parameters are evaluated (similarly to the PERFECT assessment scheme, above), such as the PFMs' endurance, repetitions, fast PFM contractions and the involuntary contraction of the PFM on coughing.
Australian Pelvic Floor Questionnaire (APFQ) | At baseline (0 week), and at the end of the intervention (12 weeks)
  Patient-centered questionnaire which assesses 42 questions in 4 domains: bladder (1-15 question), bowel ( 16-27 question), pelvic organ prolapsed (28-32 question) and sexual function (33-42 question).The scores within each domain are divided by the number of relevant questions and multiplied by 10; thus, the scores range from 0 to 10 for each domain, giving a total score from 0 to 40 (2 questions are not evaluated in the total score). Higher score indicates more severe symptoms.
Patient Global Impression of Improvement (PGI-I Scale) | At the end of the intervention (12 weeks)
  Patient-centered questionnaire where patients rate the extent to which they believe they have improved (from 1 'much better' to 7 'much worse')
Adherence questionnaire | At the middle (6 weeks), and at the end of the intervention (12 weeks)
  Patient-centered questionnaire which contains 28 questions in total and the majority of them are closed type (yes/no). The 26 questions are based on the guidelines of the World Health Organization, are divided into the following sections: a) social and demographic factors (1 to 4 questions), b) therapy-related factors (5 to 9 questions) c) healthcare team and system-related factors (physical therapists) (10 to 12 questions), d) patient-related factors (13 to 23 questions) and e) condition-related factors (24 to 26 questions). The 27 and 28 questions are related to treatment adherence. Question 27 is a 10-point scale of adherence, where patient self-assessed how well he followed the home exercise program (0-2 represent low adherence, 3-7 moderate adherence and 8-10 high adherence). Question 28 is an open-ended question about adherence to PFM exercises, where each patient explains the reason that rated himself with low or moderate adherence to the exercises.
PFM adherence exercise diary | At baseline (0 week) is provided the PFM adherence exercise diary and the patients will return it, at the end (12 weeks) of the intervention
  Patient-centered diary in which, patients fill in the daily and weekly frequency executing the PFM exersises, the sets, the repetitions and the resting periods that they folow during their treatment. If it is needed, there is a space in the diary where patients could write comments and other related infomation about the treatment prosedure.

OTHER OUTCOMES:
3-day bladder diary | At baseline (0 week) is provided the 3-day bladder diary and the patients will return it, after the 1st week
  Patient-centered diary in which, the patients fill in (during three continuous days) : (a) their daily number of incontinence incidents, (b) the daily fluid volumes (water etc) that they receive and (c) the daily quantity that they urinate.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, PhD, Study Director — University of Patras, Department of Physiotherapy
Locations (1):
- Laboratory of Clinical Rehabilitation and Research (CPRlab), University of Patras, Pátrai, Achaia, Greece

REFERENCES:
- [Background] Papanikolaou DT, Lampropoulou S, Giannitsas K, Skoura A, Fousekis K, Billis E. Pelvic floor muscle training: Novel versus traditional remote rehabilitation methods. A systematic review and meta-analysis on their effectiveness for women with urinary incontinence. Neurourol Urodyn. 2023 Apr;42(4):856-874. doi: 10.1002/nau.25150. Epub 2023 Feb 18. PMID 36808744